CLINICAL TRIAL: NCT00055120
Title: A Phase IV Study of Antiretroviral Therapy for HIV Infected Adults Presenting With Acute Opportunistic Infections: Immediate Versus Deferred Initiation of Antiretroviral Therapy
Brief Title: When to Start Anti-HIV Drugs in Patients With Opportunistic Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACTG A5164; DAIDS-ES ID 10005
Record Dates: First submitted 2003-02-19; First posted 2003-02-20 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: HIV Infections; AIDS-Related Opportunistic Infections
Keywords: Anti-HIV Agents; Disease Progression; Drug Administration Schedule; Viral Load; HIV-1; Treatment Outcome; Survival Analysis; Treatment Naive
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Disease Progression | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir; Stavudine

INTERVENTIONS:
Drug: Emtricitabine/tenofovir disoproxil fumarate
Drug: Lopinavir/ritonavir
Drug: Stavudine

SUMMARY:
The purpose of this study is to evaluate the effect of starting anti-HIV drugs in HIV infected patients who are being treated for opportunistic infections (OIs). This study will follow two patient groups: those who received anti-HIV drugs soon after being diagnosed with an OI and patients with OIs who deferred beginning anti-HIV drugs until after recovering from the OI.

DETAILED DESCRIPTION:
Despite the advent of highly active antiretroviral therapy (HAART), many HIV infected patients without access to antiretroviral therapy (ART) present with acute OIs. Such presentations pose a management problem, as there are currently no data available as to whether initiating HAART during the acute presentation is of benefit. Reports of an immune reconstitution inflammatory syndrome (IRIS) marked by increasing hypoxia or new pulmonary infiltrates have been associated with the initiation of ART in patients with AIDS. There is also concern as to drug interactions between ART and antimicrobials used to treat the presenting OI. This study will evaluate the possible benefits and costs of initiating ART in HIV infected patients who present with an AIDS-defining OI.

There are 2 steps in this study. In Step 1, patients will be randomly assigned to one of two study arms. Arm A will receive ART within 2 weeks of starting therapy for the acute OI. Arm B will have ART deferred until Step 2, at least 4 weeks and no more than 32 weeks after beginning therapy for the acute OI. Only Arm B participants will enter Step 2, which will likely begin between Weeks 6 and 12. The study will make the following drugs available for construction of an antiretroviral (ARV) regimen: emtricitabine/tenofovir disoproxil fumarate (FTC/TDF), lopinavir/ritonavir (LPV/RTV), and stavudine (d4T). Use of other ARV drugs is at the discretion of the study official. Drug regimen additions and substitutions will be made on a case-by-case basis.

Patients will be followed for 48 weeks and will have 10 study visits. All study visits will include a physical exam, medication history, and blood collection. Patients will be asked to complete questionnaires assessing health status and adherence at selected visits.

ELIGIBILITY:
Note: Participants who enrolled in this study prior to Version 3.0 will be offered and allowed to switch to FTC/TDF if they wish. However, participants under the age of 18 cannot receive FTC/TDF through this study.

Inclusion Criteria for Step 1:

* HIV-1 infected
* Currently being treated for OI (including Pneumocystis carinii pneumonia [PCP]; cryptococcal meningitis; disseminated histoplasmosis; disseminated Mycobacterium avium complex [MAC]; cytomegalovirus [CMV] retinitis; CMV encephalitis; toxoplasmic encephalitis; other atypical non-tuberculous, non-MAC mycobacterial infections; or other serious, invasive BIs). Participants who have tuberculosis (TB) alone are ineligible for this study. Participants with bacterial pneumonia or serious BI must have a CD4 count less than 200 cells/mm3 within 30 days prior to study entry. Participants with other serious OIs, including other AIDS-defining and -related OIs for which appropriate therapy other than ART exists are eligible, pending investigator approval. Participants' current OI treatment must have been started within 14 days prior to study entry, but may have been discontinued prior to study entry.
* Able to take oral medications
* Parent or guardian willing to provide informed consent, if applicable
* Willing to use acceptable methods of contraception

Exclusion Criteria for Step 1:

* Any ART within 8 weeks prior to study entry
* 31 or more days of any ARV within 6 months prior to entry
* History of more than one virologic, immunologic, or clinical treatment failure while on a HAART regimen, or a history of more than one regimen change for unknown reasons
* Systemic cancer chemotherapy within 30 days prior to study entry
* Immunomodulators within 30 days prior to study entry, including growth factors, immune globulin, interleukins, and interferons (unless for hepatitis C virus or Kaposi's sarcoma)
* Investigational ARV agents at study entry
* Systemic investigational agents (except ARV drugs) within 30 days prior to study entry will be allowed at the study official's discretion
* Anticipated use of certain medications
* Kidney failure requiring dialysis
* Current drug or alcohol use that, in the opinion of the study official, would interfere with the study
* Treatment for current, first-treated, and diagnosed OI or BI for more than 14 days prior to study entry
* Known resistance to ART that prohibits administration of an effective ART regimen
* Current OI has recurred within 90 days prior to study entry. Recurrent BIs are not excluded.
* Pregnant or breastfeeding

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2003-03; Primary Completion 2006-09 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Survival, recurrence of presenting OI/bacterial infection (BI) or incidence of new AIDS-defining events, and HIV-1 plasma viral load at Week 48

SECONDARY OUTCOMES:
HIV-1 plasma viral load at all timepoints up to and including Week 48
CD4 counts at all timepoints up to and including Week 48
changes in ARV regimen for lack of efficacy
efficacy of treatment and clinical outcomes for specific OI/BI, including duration of and complications of treatment, incidence and duration of hospitalization, rate of relapse/recurrence, and incidence of IRIS and impact on outcomes in the two arms
safety and tolerability, measured by Grade 3 and 4 signs and symptoms and laboratory toxicities, ART and OI/BI treatment changes and dose modifications due to toxicities, and IRIS
HIV-1 drug resistance over time (genotype)
health care resource use, including total inpatient days and emergency room visits compared in the two groups
quality of life (QOL) and functional status outcomes, including overall self-reported QOL and functional status compared in the two groups at Week 48
adherence, including self-reported adherence to all ARVs over the study period, examined for relationship with primary study outcomes, including death, progression, and viral suppression

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R. Zolopa, MD, Study Chair — Division of Infectious Diseases, Stanford University
Locations (45):
- United States (43):
  - University of California, Davis Medical Center, Sacramento, California
  - University of California, San Diego Antiviral Rese, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - San Mateo County AIDS Program, Stanford, California
  - Santa Clara Valley Medical Center, Stanford, California
  - Stanford Univ, Stanford, California
  - Willow Clinic, Stanford, California
  - Harbor General/UCLA, Torrance, California
  - University of Colorado Health Sciences Center, Denver, Denver, Colorado
  - Univ of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Cook County Hospital Core Center, Chicago, Illinois
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - Indiana University Hosp, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard (Massachusetts General Hospital), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Hennepin County Medical Clinic, Minneapolis, Minnesota
  - St. Louis Connect Care, St Louis, Missouri
  - Washington University (St. Louis), St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - NYU/Bellevue, New York, New York
  - Columbia University, New York, New York
  - Community Health Network, Inc., Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Presbyterian Medical Center - University of PA, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Comprehensive Care Clinic, Nashville, Tennessee
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - Univ of Texas, Galveston, Galveston, Texas
  - University of Washington (Seattle), Seattle, Washington
- University of Puerto Rico, San Juan, Puerto Rico
- University of Witwatersrand, Parktown, Johannesburg, South Africa

REFERENCES:
- [Background] Wislez M, Bergot E, Antoine M, Parrot A, Carette MF, Mayaud C, Cadranel J. Acute respiratory failure following HAART introduction in patients treated for Pneumocystis carinii pneumonia. Am J Respir Crit Care Med. 2001 Sep 1;164(5):847-51. doi: 10.1164/ajrccm.164.5.2007034. PMID 11549544
- [Background] Bartlett JA, DeMasi R, Quinn J, Moxham C, Rousseau F. Overview of the effectiveness of triple combination therapy in antiretroviral-naive HIV-1 infected adults. AIDS. 2001 Jul 27;15(11):1369-77. doi: 10.1097/00002030-200107270-00006. PMID 11504958
- [Background] Hamill RJ. Immune restoration syndrome in AIDS and mycoses. Program and abstracts of the 41st Interscience Conference on Antimicrobial Agents and Chemotherapy; December 16-19, 2001; Chicago, IL. Abtract 1272.
- [Background] Nunez M, Asencio R, Valencia ME, Leal M, Gonzalez-Lahoz J, Soriano V. Rate, causes, and clinical implications of presenting with low CD4+ cell counts in the era of highly active antiretroviral therapy. AIDS Res Hum Retroviruses. 2003 May;19(5):363-8. doi: 10.1089/088922203765551719. PMID 12803995
- [Result] Sax PE, Sloan CE, Schackman BR, Grant PM, Rong J, Zolopa AR, Powderly W, Losina E, Freedberg KA; Cepac US And Actg A5164 Investigators. Early antiretroviral therapy for patients with acute aids-related opportunistic infections: a cost-effectiveness analysis of ACTG A5164. HIV Clin Trials. 2010 Sep-Oct;11(5):248-59. doi: 10.1310/hct1105-248. PMID 21126955
- [Derived] Grant PM, Komarow L, Andersen J, Sereti I, Pahwa S, Lederman MM, Eron J, Sanne I, Powderly W, Hogg E, Suckow C, Zolopa A. Risk factor analyses for immune reconstitution inflammatory syndrome in a randomized study of early vs. deferred ART during an opportunistic infection. PLoS One. 2010 Jul 1;5(7):e11416. doi: 10.1371/journal.pone.0011416. PMID 20617176
- [Derived] Zolopa A, Andersen J, Powderly W, Sanchez A, Sanne I, Suckow C, Hogg E, Komarow L. Early antiretroviral therapy reduces AIDS progression/death in individuals with acute opportunistic infections: a multicenter randomized strategy trial. PLoS One. 2009;4(5):e5575. doi: 10.1371/journal.pone.0005575. Epub 2009 May 18. PMID 19440326